CLINICAL TRIAL: NCT06396013
Title: A Multicentre Randomized Controlled Clinical Study on the Chitosan Nanocrystalline Qinteng Huoxue Runji Ointment Therapy for Psoriasis With Blood Stasis Syndrome.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Liyun Sun, chief physician, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: shoufa2024-2-2237
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Plaque Psoriasis
Keywords: Plaque psoriasis; blood stasis syndrome; Qinteng Huoxue Runji Ointment; chitosan; randomized controlled trial
MeSH Terms: interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group received topical Chitosan Nanocrystalline Qinteng Huoxue Runji Ointment, twice a day for 12 weeks
  Interventions: Drug: Chitosan Nanocrystalline Qinteng Huoxue Runji Ointment
- control group (Placebo Comparator): The control group received topical placebo twice a day for 12 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Chitosan Nanocrystalline Qinteng Huoxue Runji Ointment — Basic treatment: According to the recommendations of the Guidelines, all participant took the traditional Chinese medicine decoction Huoxue Sanyu Decoction orally. 2 times/day for 12 weeks.
  Acute administration: When the participant has unbearable itching, the doctor can give loratadine tablet 10mg orally once a night, and record the dosage and frequency of use.
  Other Names: TCM decoction Huoxue Sanyu Decoction; Loratadine
  Arms: experimental group
Drug: placebo — Basic treatment: According to the recommendations of the Guidelines, all participant took the traditional Chinese medicine decoction Huoxue Sanyu Decoction orally. 2 times/day for 12 weeks.
  Acute administration: When the participant has unbearable itching, the doctor can give loratadine tablet 10mg orally once a night, and record the dosage and frequency of use.
  Other Names: Loratadine
  Arms: control group

SUMMARY:
Background: Psoriasis is one of the hot spots in the field of skin disease prevention and treatment, and TCM topical preparations have unique advantages in the treatment of psoriasis. The Qinteng Huoxue prescription series of TCM topical preparations created by Professor Sun Liyun have been observed to be effective in clinical practice in the treatment of psoriasis, but there is no multi-center clinical trial for blood stasis syndrome. In addition, the TCM topical preparations has the disadvantages of large particle diameter and unfavorable penetration of skin barrier.

Objective: In this study, chitosan nanocrystalline drug delivery system was used to prepare Chitosan Nanocrystalline Qinteng Huoxue Runji Ointment, and the efficacy and safety of Chitosan Nanocrystalline Qinteng Huoxue Runji Ointment in the intervention of psoriasis with blood stasis syndrome was investigated through multi-center, randomized, double-blind, self-controlled bilateral skin lesions and placebo-controlled clinical trials.

Methods: A total of 96 patients with plaque psoriasis with blood stasis syndrome of were enrolled in 4 research centers, and bilateral symmetrical rashes on limbs or trunk were selected, and randomly divided into experimental group and control group. The experimental group received topical Chitosan Nanocrystalline Qinteng Huoxue Runji Ointment, twice a day for 12 weeks, and the control group received topical placebo twice a day for 12 weeks, and two follow-up visits were performed at the 16th and 20th week.

Results Indicators: The main efficacy indicators were targeted psoriasis area and severity index (tPASI), and the secondary efficacy indicators included: Psoriasis physician global assessment (PGA), target lesion area, numerical rating scale (NRS), TCM syndrome score, dermatology life quality index (DLQI), MOS 36 item short from health survey (SF-36)), and the morphology and number of vascular globules under dermoscopy. tPASI, PGA, target lesion area, NRS were assessed at baseline, at 2, 4, 6, 8, 10, 12 weeks of treatment, and at 16 and 20 weeks of follow-up. TCM syndrome score, DLQI, SF-36, and dermoscopy were assessed at baseline, 12 and 20 weeks. Safety assessment includes vital signs monitoring, blood routine, urine routine, liver and kidney function tests, and adverse events and adverse reactions. SPSS 20.0 was used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria of plaque psoriasis vulgaris;
2. Meets the diagnostic criteria of plaque psoriasis with blood stasis syndrom;
3. 18 ≤ age ≤65 , gender is not limited;
4. Quiescent patients;
5. Severity of the disease: mild to moderate lesions were 3≤PASI≤10, and 3≤BSA≤10;
6. Volunteers can understand the research content and sign the informed consent voluntarily. The informed consent process complies with the provisions of the GCP.

Exclusion Criteria:

1. psoriasis induced by drug factors; Combined with non-plaque psoriasis (i.e. guttate, joint, pustule, erythroderma, or other types of psoriasis); Skin lesions were found only in special parts of the face, scalp, nails, creases, glans, mucous membranes, palms and plantar.
2. Received abiotic agents of systemic drug therapy within 4 weeks prior to randomization, including but not limited to systemic glucocorticoids, retinoids, methotrexate, and cyclosporine;
3. Received biologics within 12 weeks or 5 half-lives prior to randomization (whatever is longer), including but not limited to interleukin antibodies (e.g. Usinumab, secuchiumab, etc.) and tumor necrosis factor a antagonists (e.g. Etanercepp, infliximab, adalimumab, etc.);
4. Local topical psoriasis treatment, including retinoids, vitamin D3 derivatives, glucocorticoids, etc., had been received within 2 weeks before randomization;
5. Use of physical therapy within 4 weeks before randomization, including phototherapy (such as UVB, PUVA), phototherapy combined therapy, bath therapy, etc.;
6. systemic anti-infection therapy within 4 weeks prior to randomization; A recurrent, chronic, or active infection at baseline that the investigator determined would increase the subject's risk;
7. with a serious, progressive, or uncontrolled disease, including but not limited to past or current autoimmune disease (such as: Rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, etc.) or diseases of the endocrine system, blood system, urinary system, hepatobiliary system, respiratory system, nervous system, mental system, cardiovascular system, gastrointestinal system or infectious diseases, malignant tumors; A history of drug abuse, alcohol/drug abuse;
8. Patients with serum creatinine higher than the upper limit of normal, glutamic pyruvic transaminase or glutamic oxalacetic transaminase level ≥1.5 times the upper limit of normal;
9. Patients who have participated in clinical trials and used investigational drugs within 1 month;
10. Patients who are allergic to known components of the trial intervention;
11. The patient (including the partner) has a pregnancy plan from 2 weeks before the first dose to 1 month after the last dose or is unwilling to take effective contraceptive measures during pregnancy or lactation;
12. There are circumstances that other investigators consider unsuitable for study participation, such as subjects with other skin problems that hinder the evaluation of psoriasis, potential compliance problems, inability to complete all examinations and evaluations as required by the protocol, and uncontrollable risks to study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
tPASI | week0 2 4 6 8 10 12 16 20
  targeted psoriasis area and severity index

SECONDARY OUTCOMES:
PGA | week0 2 4 6 8 10 12 16 20
  physician global assessment
target lesion area | week0 2 4 6 8 10 12 16 20
  target lesion area
NRS | week0 2 4 6 8 10 12 16 20
  numerical rating scale
TCM syndrome score | week0 12 20
  TCM syndrome score
DLQI | week0 12 20
  dermatology life quality index
SF-36 | week0 12 20
  MOS 36 item short from health survey
the morphology and number of vascular globules under dermoscopy | week0 12 20
  the morphology and number of vascular globules under dermoscopy

IPD SHARING:
Plan to Share IPD: No